CLINICAL TRIAL: NCT00099827
Title: Teen Depression Awareness Project- This Project Examines the Services Used by Teens Identified in Primary Care Settings With Depression
Brief Title: Teen Depression Awareness Project (TDAP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Audrey Burnam, RAND
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TDAP2
Record Dates: First submitted 2004-12-21; First posted 2004-12-21 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Education — Individuals will receive information about depression

SUMMARY:
The main objective of this research project is to describe the impact of depression on adolescent and family functioning compared to that of healthy adolescents and to understand the impact of Feedback and Patient Activation (FPA) on teen and family decision-making regarding seeking care for depressive disorders.

DETAILED DESCRIPTION:
Background: Depressive disorders are common among adolescents, and efficacious treatments are available. However, few adolescents receive appropriate care, and the effects of these disorders on adolescents' functioning and family burden are not well understood. Documenting these effects could make identifying and treating adolescents with mental health problems a higher priority for providers and parents, and for the adolescents themselves, than it is now.

Primary care settings provide the most important opportunities to improve care for mood and anxiety disorders among adolescents, since most children and adolescents have some contact with a primary care provider each year for well-child visits, school physicals, or acute care. However, an ongoing trial of a quality improvement intervention for depressed adolescents in primary care settings (RAND's Youth Partners in Care study) suggests that there are significant barriers to implementing quality improvement protocols in primary care.

Study Goals: The main objective of this research is to build an empirical foundation for developing effective strategies to improve treatment of adolescent mood and anxiety disorders in primary care settings. Our specific goals are to:

1. Describe the impact of depression on adolescent and family functioning compared to that of healthy adolescents.
2. Evaluate the effect of two interventions--depression diagnosis feedback and an educational brochure, with or without patient activation, on care received.
3. Identify barriers and facilitators to receiving appropriate care for identified adolescent depression from the perspective of adolescents, parents, and the primary care providers.

Methodology: Participants for this study will be recruited from three to four study sites in each of two cities selected from among eligible general health care settings that serve high volumes of adolescent patients, including a large community-based clinic and a set of small clinics; a high school-based health clinic; and a public/free clinic.

Specific aim 1: We will describe the impact of depression on adolescent and family functioning compared to healthy controls using a 2-group longitudinal comparison between 400 adolescents identified at baseline with major depression, and 400 adolescents with no detectable mental disorders. Primary data will be collected from three types of respondents: adolescents aged 13-17, their parents, and their health care providers. Adolescent baseline and follow-up assessments (for behavioral problems, physical health, health-related quality of life, use of psychotropic medications, etc.) will be conducted through telephone interviews supplemented by mailed questionnaires. Parents will be asked to complete baseline and follow-up assessments to determine family burden, health insurance, demographics, and the adolescent's functioning at school. Study participants will be assessed twice, 6 months apart, with an interim contact at 3 months. Primary care providers (PCPs) will complete written questionnaires that will include data on demographic characteristics, medical background and training, professional practices, as well as knowledge, attitudes and reported treatment behaviors.

Specific aim 2: We will evaluate the effect of the intervention on care received by randomizing half of the 400 adolescents with major depression to one of two conditions--Feedback and Educational Brochure, with and without Patient Activation (FPA) and then observing service use over the next 6 months. The minimal intervention consists of feedback about the diagnosis to the primary care provider, teen and parent, and also includes an educational brochure to teens and parents. In the more active FPA intervention, in addition to feedback and educational brochure, telephone calls will be made to depressed teens and their parents to discuss symptoms and alternative treatment options with the aim of encouraging help-seeking. We will compare the two groups on whether they received mental health care, what kind, and their satisfaction with that care.

Specific aim 3: For the 400 depressed teens in the study, we will conduct a descriptive analysis of the preferences for treatment, barriers encountered, and use of services. We will obtain this information from the teens', parents', and providers' perspectives in order to identify barriers and facilitators to receiving appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 13-17
* Attending School
* Living with parent or guardian
* Reads and writes English
* Receiving care at a participating PCP office

Exclusion Criteria:

* Pregnancy
* Parents don't speak English or Spanish

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 368 (Actual)
Dates: Start 2003-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Receipt of Care | September 30, 2007

SECONDARY OUTCOMES:
Journal Article | September, 2007
Journal Articles | September, 2007

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Burnam, PhD, Principal Investigator — RAND
Locations (8):
- United States (8):
  - Family Care Specialists at White Memorial Medical Center, Los Angeles, California
  - Northeast Valley Health Corporation-San Fernando Valley High School, San Fernando, California
  - Children's National Medical Center Adolescent Health Clinic, Washington D.C., District of Columbia
  - Children's Pediatricians and Associates, Washington D.C., District of Columbia
  - Capital Medical Group, Chevy Chase, Maryland
  - Kaiser Mid-Atlantic, Kensington, Maryland
  - Kaiser Mid-Atlantic, Rockville, Maryland
  - Kaiser Mid-Atlantic-Camp Springs, Temple Hills, Maryland